CLINICAL TRIAL: NCT02857257
Title: Transplantation of Anaerobic Cultured Human Intestinal Microbiota in Irritable Bowel Syndrome
Acronym: ACHIM2
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Uppsala University (Other)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Per Hellström, Professor, Uppsala University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACHIM2
Record Dates: First submitted 2016-07-26; First posted 2016-08-05 (Estimated); Last update posted 2018-08-08 (Actual); Status verified 2018-08

CONDITIONS: Irritable Bowel Syndrome
Keywords: IBS; Microbiota
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment arm (Experimental): Only one treatment arm. Patients are allocated under disease condition and later treated with ACHIM. The post-treatment disease progression is monitored.
  Interventions: Biological: ACHIM

INTERVENTIONS:
Biological: ACHIM — After an observation period of 4 weeks patients with IBS-D will be treated with ACHIM
  Other Names: Anaerobic cultured human intestinal microbiota

SUMMARY:
Patients with irritable bowel syndrome (IBS) are treated with microbiota from a human intestinal anaerobic sample cultured for decades. Patients are recruited consecutively with symptoms of IBS and serve as their own controls. After an observation time of 4 weeks, patients are recruited for a 1-week run-in and then given the cultured fecal microbiota by the duodenal route via gastroscopy. Two treatments are given within a 1-week interval. Assessment of symptoms are made before and 4 weeks after the last treatment (at 6 weeks). Additionally, fecal samples are collected for bacterial 16S ribosomal ribonucleic acid (rRNA) analysis and bacterial functional parameters (microflora-associated characteristics).

DETAILED DESCRIPTION:
Diarrhea-dominated irritable bowel syndrome (IBS-D) is studied in subjects by treatment with an anaerobic human intestinal microbiota cultured for 15 years and quality controlled with a specified content of bacterial species regularly over the years. Inclusion criteria is: Diarrheal disease since at least 4 weeks, 18-80 years of age, previously unsuccessful treatment with no symptomatic relief of antidiarrheals or resins, and signed informed consent.

Primary outcome was irritable bowel syndrome-symptom severity scale (IBS-SSS). Secondary outcome was Bristol stool scale (BSS).

Secondary outcome: Changes in fecal microflora distribution and multiplicity as shown by the 16S ribosomal ribonucleic acid (rRNA) analysis of feces.

Once eligible for the study, patients were monitored for a run-in period of one week with the IBS-SSS and the BSS plus fecal samples for analysis of bacterial species using the bacterial specific 16S rRNA differentiation.

Then, the anaerobic cultured human intestinal microflora (ACHIM) was given twice with an interval of 1 week. Thereafter, patients were further monitored over 4 weeks as regards IBS-SSS and BSS. Another feces sample was also collected for bacterial 16S rRNA analysis to evaluate the microbiota diversity.

The study will be evaluated using eligible subjects as their own controls by means of Wilcoxon's matched-pairs test, alternatively t-test for matched pairs.

Power analysis show that 40 subjects are needed to study in order to achieve a power of 80%.

ELIGIBILITY:
Inclusion Criteria:

* IBS according to the Rome III criteria

Exclusion Criteria:

* Pregnancy
* Antibiotic and probiotics within 8 weeks before inclusion
* Unable to give informed consent
* Immunodeficiency (drug- och disease-related)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-01; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Symptom relief according to irritable bowel syndrome-symptom severity scale (IBS-SSS) | 4 weeks

SECONDARY OUTCOMES:
Differential bacterial species population as defined by 16S RNA | 4 weeks
  Description of different bacterial species harboring in fecal samples before and after treatment with ACHIM. Exploratory outcome measure.
Normalization of stool consistency as determined by the Bristol stool scale | 4 weeks
  Normalization as determined by the Bristol stool scale

CONTACTS AND LOCATIONS:
Overall Officials: Per Hellström, MD, PhD, Study Director — Uppsala University
Locations (1):
- Mag-tarm/endoskopienheten Hötorget, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Francis CY, Morris J, Whorwell PJ. The irritable bowel severity scoring system: a simple method of monitoring irritable bowel syndrome and its progress. Aliment Pharmacol Ther. 1997 Apr;11(2):395-402. doi: 10.1046/j.1365-2036.1997.142318000.x. PMID 9146781
- [Result] Lewis SJ, Heaton KW. Stool form scale as a useful guide to intestinal transit time. Scand J Gastroenterol. 1997 Sep;32(9):920-4. doi: 10.3109/00365529709011203. PMID 9299672
- [Result] Smits LP, Bouter KE, de Vos WM, Borody TJ, Nieuwdorp M. Therapeutic potential of fecal microbiota transplantation. Gastroenterology. 2013 Nov;145(5):946-53. doi: 10.1053/j.gastro.2013.08.058. Epub 2013 Sep 7. PMID 24018052
- [Derived] Benno P, Norin E, Midtvedt T, Hellstrom PM. Therapeutic potential of an anaerobic cultured human intestinal microbiota, ACHIM, for treatment of IBS. Best Pract Res Clin Gastroenterol. 2019 Jun-Aug;40-41:101607. doi: 10.1016/j.bpg.2019.03.003. Epub 2019 Apr 29. PMID 31594647